CLINICAL TRIAL: NCT02156349
Title: Integrated Personalized Diabetes Management (Integrated PDM): Prospective, Randomized, Controlled Intervention Study for the Evaluation of the Effectiveness and the Benefit of Integrated PDM in the Care of People With Type 2 Diabetes in Diabetes Specialized Medical Practices in Germany (DSP)
Brief Title: A Study Evaluating the Efficacy and the Benefit of Integrated Personalized Diabetes Management (PDM) for Diabetic Patients.
Acronym: PDMProValueDSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD001732
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Type II Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

ARMS (2):
- Control Group (Other): Patients treated by usual customary medical practice (Usual Care) in the out-patient facility i.e. Diabetes specialized medical practice, Medical Care Center or hospital outpatient clinic.
  Interventions: Device: Accu-Chek Smart Pix readout Device
- Intervention group (Other): Patients are treated according to the concept "Integrated personalized diabetes management".
  Interventions: Device: Accu-Chek Smart Pix Software

INTERVENTIONS:
Device: Accu-Chek Smart Pix Software — Software with adherence evaluation software used according to Integrated Personalized Diabetes Management (PDM)
  Arms: Intervention group
Device: Accu-Chek Smart Pix readout Device — Smartpix device for data upload out of blood glucose meter devices
  Arms: Control Group

SUMMARY:
This study is a German, prospective, multicenter, controlled, cluster-randomized, interventional comparative study evaluating the efficacy and benefits of integrated PDM care by measuring HbA1c levels in patients with Type 2 Diabetes. Patients will be randomized into two groups to use Accu-Chek Smartpix software and Accu-Chek Smartpix device.

DETAILED DESCRIPTION:
Outcome of both studies (RD001732 and RD001231) will be integrated and additionally reported as PDM-ProValue study program (Integrated Personalized Diabetes Management) due to the high similarity in study characteristics, design and study results.

ELIGIBILITY:
Inclusion Criteria:

* existence of a signed Informed Consent form (before any study procedure)
* diagnosed Type 2 diabetes mellitus
* age ≥18 years
* insulin therapy for ≥6 months: BOT, SIT, CT or ICT
* HbA1c ≥7.5% (≥ 58,47 mmol/mol respectively), blood withdrawal for measurement in the last 90 days before study visit 1 (patient's inclusion)
* longer-term care (at least for the duration of the 12-month study participation) by the trial site
* insured by the statutory health insurance (GKV) as a compulsory member or voluntarily insured member or as a family co-insured member
* willing and able to participate in the study and to follow the study procedures, among other things sufficient command of the German language, spoken and written

Exclusion Criteria:

* Treatment of diabetes with insulin pump (CSII)
* Methodic and continuous with the use of particular software for processing of SMBG data - by the patient and at visits in the practice by the physician/diabetes educator - in the past 12 months before study participation.presence of terminal renal failure (eGFR < 15ml/min) / dialysis and/or a loss of sight (visual acuity ≤ 0,05 of the better eye)
* Existing tumor illness (primary tumor/local recurrence/ metastases except Basal Cell Carcinoma) in the past 5 years before study participation newly diagnosed or treated acutely (hormone, chemo- or radiation therapy). Within a tumor free time of < 5 years Medical Affairs will decide about individual cases
* permanent use of steroids in adrenal suppressant doses, of other immuno-modulatory drugs or chemotherapy
* known alcohol and drug abuse and medication abuse
* known metabolic disorders and/or disorders or therapies that could lead to or have led to wrong measured results (e.g. with the blood glucose measurement)
* existing pregnancy, breast-feeding or plan to become pregnant during study participation
* physical illness and/or psychological disorder with the result that the patient cannot implement the medical treatment recommendations independently
* dependency relationship to the sponsor or to the investigator, e.g. as a professional colleague or family member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
The mean HbA1c change by means of Generalized Estimating Equations (GEE) methods | from Baseline to 12 months
  The difference in the HbA1c change after 12 months between the Intervention group and the Control group is analyzed by means of generalized estimating equations (Generalized Estimating Equations [GEE]) methods (population averaged model) and here, robust assessors (so-called sandwich assessors) for the standard errors are provided. The dependent variable is the HbA1c change after 12 months, while the HbA1c baseline considers the gender and the age as factors of influence (covariates) in the GEE model.

SECONDARY OUTCOMES:
Effects of integrated Personalized Diabetes Management (PDM) by means of Generalized Estimating Equations [GEE] methods | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Iris Vesper, Study Director — Roche Diabetes Care
Locations (50):
- Germany (50):
  - Private Practice, Altenstadt
  - Internistische Gemeinschaftspraxis, Augsburg
  - Forschungsinstitut der Diabetes Akademie Mergentheim (FIDAM), Bad Mergentheim
  - Private Practice, Bad Säckingen
  - Private Practice, Berlin
  - MVZ am Bahnhof Spandau, Berlin
  - Gemeinschaftspraxis, Bitburg
  - Private Practice, Buxtehude
  - Praxis Kugler, Cologne
  - Private Practice, Cuxhaven
  - Diabetologicum Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Gemeinschaftspraxis Schaden, Düsseldorf
  - Private Practice, Essen
  - Schwerpunktpraxis für Diabetes, Gefäß- und Ernährungsmedizin, Falkensee
  - Private Practice, Frankfurt am Main
  - Gemeinschaftspraxis, Fulda
  - Private Practice, Gelnhausen
  - Hausärztliche internistische Gemeinschaftspraxis Giessen, Giessen
  - Diabetes- und Gesundheitszentrum Göttingen, Göttingen
  - Private Practice, Gummersbach
  - Private Practice, Hamburg
  - Diabeteszentrum, Hamburg
  - Private Practice, Hanau
  - Integriertes Diabetiker-Zentrum Hannover, Hanover
  - Gemeinschaftspraxis, Herne
  - Gemeinschaftspraxis im Altstadt-Carree, Hessen
  - Private Practice, Immenhausen
  - Universitätsklinikum Jena, Klinik für Innere Medizin III, Jena
  - Diabeteszentrum Kassel, Kassel
  - Internistische Praxis Lampertheim, Lampertheim
  - Private Practice, Lauf (Pegnitz)
  - Private Practice, Laupheim
  - Private Practice, Lingen
  - Diabetes-Zentrum Neustadt, Neustadt am Rübenberge
  - Diabetologische Schwerpunktpraxis, Nordrhein-Westfalen
  - Private Practice, Offenbach
  - Diabetes Praxis Oranienburg, Oranienburg
  - Arztpraxis fur Allg-Med, Pirna
  - Private Practice, Porta Westfalica
  - Private Practice, Rehburg-Loccum
  - Gemeinschaftspraxis, Rhaunen
  - Pivate Practice, Rüsselsheim am Main
  - Ambulanzzentrum Schweinfurt, Schweinfurt
  - Versdias Gmbh, Sulzbach-Rosenberg
  - Private Practice, Trier
  - Gemeinschaftspraxis am Bärenplatz, Villingen-Schwenningen
  - Diabetolog. Schwerpunktpraxis, Wiesbaden
  - Internistische Praxis, Zierenberg
  - Arztpraxis Zossen / Dabendorf, Zossen